CLINICAL TRIAL: NCT02036632
Title: Eye Patching as a Potential Treatment Modality for and a Possible Etiological Insight on Central Serous Retinopathy
Brief Title: Eye Patch Therapy for Central Serous Retinopathy (CSR)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201211016
Record Dates: First submitted 2014-01-08; First posted 2014-01-15 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Central Serous Retinopathy (CSR)
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eye Patching (Other): Intervention
  Interventions: Device: Eye Patching

INTERVENTIONS:
Device: Eye Patching

SUMMARY:
First, this study will investigate the viability of 24-hour eye patching as a potential treatment modality for CSR. Second, this study will assess a potential physiologic explanation for CSR, namely if inhibition of photic stimulation of the diseased retina will aid in ameliorating disease severity and disease duration.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older
* Both males and females
* Patients diagnosed with active central serous retinopathy
* Patients who are willing to use an eye patch in the affected eye for 24 hours
* Patients who are able to make the follow up appointments as required by the study

Exclusion Criteria:

* Individuals under 18 years of age
* Patients with vision less than 20/40 in the unaffected eye.
* Patients who are not able to undergo mfERG testing in a realiable manner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in multi-focal ERG response and macular thickness after 24-hour patch therapy in patients with CSR | 24 hours
  This study is a prospective control trial that will compare 24-hour eye patch therapy with the current standard of care in patients with central serous retinopathy (CSR).
Change in multi-focal ERG response | 24 hours

SECONDARY OUTCOMES:
macular thickness | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P Van Stavern, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington Universtiy School of Medicine, St Louis, Missouri, United States